CLINICAL TRIAL: NCT00595660
Title: Best Needle Size for FNA of Palpable Breast Mass:Randomised Controlled Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kashani Social Security Hospital (Other)
Responsible Party: Dr.Hamidzadeh, Kashani Social Security Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 17251-10/10/1386
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Last update posted 2008-01-16 (Estimated); Status verified 2008-01

CONDITIONS: Palpable Breast Mass
Keywords: Palpable Breast Mass; FNA; Cytology; Fine needle aspiration; Specimen Adequacy
MeSH Terms: interventions — Biopsy, Fine-Needle

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): Needle 21 for FNA
  Interventions: Procedure: FNA - fine needle aspiration
- 2 (Active Comparator): 22 needle for FNA
  Interventions: Procedure: FNA - fine needle aspiration
- 3 (Active Comparator): 23 needle for FNA
  Interventions: Procedure: FNA - fine needle aspiration
- 4 (Active Comparator): 24 needle for FNA
  Interventions: Procedure: FNA - fine needle aspiration

INTERVENTIONS:
Procedure: FNA - fine needle aspiration — Fine Needle aspiration
Procedure: FNA - fine needle aspiration — Fine needle aspiration
  Arms: 1
Procedure: FNA - fine needle aspiration — Fine needle aspiration
  Arms: 2
Procedure: FNA - fine needle aspiration — Fine needle aspiration
  Arms: 3
Procedure: FNA - fine needle aspiration — Fine needle aspiration
  Arms: 4

SUMMARY:
Needle size from22 to 25 were used for fine needle aspiration of palpable breast lumps. In this study we choose one, randomly, and fallow the result of cytologic evaluation regarding specimen adequacy.

DETAILED DESCRIPTION:
Patient assigned randomly to FNA of palpable breast mass with different needle size:21-22-23-24

ELIGIBILITY:
Inclusion Criteria:

* Any Woman with palpable Breast Mass

Exclusion Criteria:

* Previous open Biopsy or Surgery
* Active infection
* Breast cysts
* Patient refusal to do FNA

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2008-02; Primary Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
specimen adequacy | 2 years

SECONDARY OUTCOMES:
complication | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bijan Mohammadhosseini, General Surgeon,MD, Principal Investigator — Kashani Social Security Hospital
Locations (1):
- Kashani Social Security Hospital, Tehran, Tehran Province, Iran